CLINICAL TRIAL: NCT02001870
Title: Comparison of the Efficiency of Intra-uterine Insemination and in Vitro Fertilization in Women Over 37 Years
Acronym: AMPAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recuitment target non obtained
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/12/0553; National PHRC 2012 (Other Grant/Funding Number: Ministère des affaires sociales et de la santé)
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Infertilities
Keywords: Infertility; female age; intra-uterine insemination; in vitro fecundation; assisted reproductive technology center
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In Vitro Fecundation (IVF) (Experimental): Couples will be treated by In Vitro Fecundation (IVF)
  Interventions: Procedure: In Vitro Fecundation (IVF)
- Intra Uterine Insemination (IUI) (Active Comparator): Couples will be treated by Intra Uterine Insemination (IUI)
  Interventions: Procedure: Intra Uterine Insemination (IUI)

INTERVENTIONS:
Procedure: In Vitro Fecundation (IVF) — In vivo fertilization will be performed according to the usual procedure of each Assisted Reproductive Technology (ART) center.
  Arms: In Vitro Fecundation (IVF)
Procedure: Intra Uterine Insemination (IUI) — Intra-uterine insemination will be performed according to the usual procedure of each ART center
  Arms: Intra Uterine Insemination (IUI)

SUMMARY:
As age increases the chances for a woman to become pregnant decrease as well spontaneously as through assisted reproductive technologies (ART). For the treatment of unexplained infertilities two techniques can be used: intra-uterine insemination (IUI) and in vitro fertilization (IVF). The aim of the present study is to compare the efficiency in term of delivery rate of IUI and IVF in couples in whom the female age is over 37 years.

DETAILED DESCRIPTION:
IUI can be used to treat infertility when tubes are normal, with no severe endometriosis and enough motile spermatozoa can be inseminated. In these cases IUI are usually performed (4 to 6 attempts) and IVF only in case of IUI failure. Indeed if the pregnancy rate per attempt is higher with IVF, IUI can be performed more frequently (6 times a year vs. 2 for IVF) so that the pregnancy rates after one year of treatment are close. When female age is over 37 years, some ART centers prefer to perform directly IVF, since chances of pregnancy decreases with time. However there is no argument in the literature in favor as well as in disfavor for such an attitude. Indeed the delivery rates after one year treatment with IUI or IVF are not known in this population. Therefore we propose a multicentric randomized controlled trial comparing IUI and IVF in women over 37 with unexplained infertility. Couples will be randomly allocated to IUI or IVF during one year. In case of absence of pregnancy after 4 IUI, couples will be treated by IVF. ART attempts will be performed according to usual procedures of each center. The follow-up will be ended either at the end of the first year of treatment if no pregnancy is obtained or at the time of delivery if a pregnancy is obtained. All data of attempts (demographics data, type and doses of treatment, adverse effects, outcome, number and health state of newborns....) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 37 and 42 years at the time of inclusion
* Infertility duration ≥ 12 months
* Normal tubes
* No severe endometriosis
* At least 1.5 106 motile spermatozoa to be inseminated
* No previous ART attempt

Exclusion Criteria:

* Tubal abnormalities
* Severe endometriosis
* Less than 1.5 106 motile spermatozoa to be inseminated
* Use of frozen sperm
* Presence of anti-spermatozoa antibodies

Ages: 37 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Delivery rate. | After one year of treatment.

SECONDARY OUTCOMES:
Multiple pregnancy rate | After one year of treatment.
Cost of treatment | After one year of treatment.
Adverse effects (hyperstimulation, infections…) | After one year of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean PARINAUD, MD, Principal Investigator — University Hospital of Toulouse
Locations (12):
- France (12):
  - University Hospital, Toulouse, Midi-Pyrénnées
  - CHU Bordeaux Hôpital Pellegrin, Bordeaux
  - CHRU Brest Hôpital Morvan, service d'AMP, Brest
  - Centre Hospitalier Intercommunal de Créteil, Service d'AMP, Créteil
  - CHU Dijon Laboratoire de biologie de la reproduction, Dijon
  - Institut de Médecine de la Reproduction, Marseille
  - CHU Montpellier, Médecine de la Reproduction, Montpellier
  - CHU Nantes centre d'AMP, Nantes
  - CHU Nice centre d'AMP, Nice
  - CHI Poissy St-Germain en Laye, centre d'AMP, Poissy
  - Centre Hospitalier des Quatre Villes, Saint-Cloud Service de Médecine de la Reproduction, Saint-Cloud
  - CHU de Strasbourg, Centre d'AMP, Strasbourg